CLINICAL TRIAL: NCT00088504
Title: A Phase 2b Study of Merimepodib in Combination With Pegylated Interferon Alfa-2a (Pegasys®) and Ribavirin in Subjects With Chronic Hepatitis C Non-Responsive to Prior Therapy With Pegylated Interferon Alfa and Ribavirin
Brief Title: Merimepodib (MMPD) in Triple Combination for the Treatment of Chronic Hepatitis C
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Robert Kauffman, M.D., Ph.D., Vertex Pharmaceuticals Incorporated
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VX03-497-205
Record Dates: First submitted 2004-07-27; First posted 2004-07-28 (Estimated); Last update posted 2007-12-21 (Estimated); Status verified 2007-12

CONDITIONS: Hepatitis C; Hepatitis
Keywords: Hepatitis
MeSH Terms: conditions — Hepatitis C; Hepatitis | interventions — N-3-(3-(3-methoxy-4-oxazol-5-ylphenyl)ureido)benzylcarbamic acid tetrahydrofuran-3-yl ester; peginterferon alfa-2a; Ribavirin

INTERVENTIONS:
Drug: Merimepodib
Drug: PEG-Interferon-alpha 2a (Pegasys®)
Drug: Ribavirin (Copegus®)

SUMMARY:
This trial is designed to test whether or not the addition of merimepodib (MMPD) to the standard therapy of pegylated interferon and ribavirin will result in a positive treatment response for people who have not previously responded to this therapy. Approximately 315 subjects will be enrolled in this research study at approximately 55 clinical sites in the United States. There will be three study groups. Everyone in the study will receive Pegasys® (pegylated interferon) and Copegus® (ribavirin) at the normally prescribed doses. Two of the groups will also receive the study drug merimepodib (MMPD) twice a day, one group at each dose level being tested. The third group will take a placebo instead of MMPD, with the Pegasys® and Copegus®.

After the first 24 weeks of treatment, blood tests will be done to see if subjects are responding to treatment. If they are responding, they will continue receiving study treatment in the study for another 24 weeks. If they are not responding, they will stop study treatment. Everyone who is responding will be monitored for 24 weeks after the last dose of medication, to see how long the response lasts.

Evaluations will be performed during the study to look at the safety of the Pegasys®/Copegus® and MMPD or placebo combination, and to see how the combination is working by measuring Hepatitis C Virus in the blood.

At some of the clinical sites performing the study, some subjects may also participate in additional testing to look at the metabolism of the drugs, or to look at the immune response to Hepatitis C virus infection and treatment.

ELIGIBILITY:
Inclusion Criteria:

The following is a summary of the inclusion and exclusion criteria for the Merimepodib Triple Combination (METRO) trial. There are also additional criteria, which will be reviewed with you by the staff at the clinical study site, to make sure you are eligible for the study. Some of the criteria are dependent on the results of blood tests and other tests that will be done at the clinical site.

If you are not sure whether you meet these criteria, please call the clinical study site nearest you, and they can help you figure out if you might be eligible for the study:

* You must have been diagnosed with Hepatitis C.
* You must have been treated with pegylated interferon (brand names are Pegasys® or Peg-Intron®) and ribavirin (brand names Rebetol® or Copegus®), for at least 12 weeks. However, you cannot have received more than one course of this combination therapy.
* You must have been a "non-responder" to this treatment, meaning that the virus levels in your blood were always detectable. If you responded to the treatment and then the virus became detectable again (called a "relapse"), you would not be eligible.
* You must not have used illegal drugs, or have a history of significant alcohol use, within the last year before you start the study.

Pegasys® and Copegus® are not recommended for people with some illnesses. You should be in good health in general, with no illnesses that would prevent you from using Pegasys® and Copegus®. If you do not know whether you have any illness or conditions that would prevent you from using these medications, the study doctor or nurse will review your medical history with you to determine this.

If you are a woman who can have children, you must be willing to use two effective methods of birth control during the study and for 6 months after the last dose of the medication. You will have monthly pregnancy tests during this time to make sure you do not become pregnant (This is recommended for anyone taking ribavirin, even when they are not in a clinical study.).

If you are a male, your female partner must not be pregnant, and you both must be willing to use birth control during the time you are in the study, and for 6 months after the last dose of the medication (This is recommended for anyone taking ribavirin, even when they are not in a clinical study.).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 315
Dates: Start 2004-07; Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Kauffman, MD, PhD, Study Director — Vertex Pharmaceuticals Incorporated
Locations (67):
- United States (67):
  - Joseph L. Cochran, M.D., Birmingham, Alabama
  - Suresh Karne, M.D., Ph.D., Huntsville, Alabama
  - Vijayan Balan, M.D., Phoenix, Arizona
  - Michael P. DeMicco, M.D., Anaheim, California
  - Prahalad B. Jajodia, M.D., Fresno, California
  - F. Fred Poordad, M.D., Los Angeles, California
  - Ramsey Cheung, M.D., Palo Alto, California
  - Myron J. Tong, M.D., Ph.D., Pasadena, California
  - Michael T. Bennett, M.D., San Diego, California
  - Lisa M. Nyberg, M.D., San Diego, California
  - Natalie Bzowej, M.D., San Francisco, California
  - Marcelo Kugelmas, M.D., Englewood, Colorado
  - Herbert L. Bonkovsky, M.D., Farmington, Connecticut
  - Eugene R. Schiff, M.D., Miami, Florida
  - Jawahar L. Taunk, M.D., Palm Harbor, Florida
  - Arnold L. Lentnek, M.D., Marietta, Georgia
  - Ellen B. Hunter, M.D., Boise, Idaho
  - Steven L. Flamm, M.D., Chicago, Illinois
  - Helen Te, M.D., Chicago, Illinois
  - Gerald J. Mingoletti, M.D., Oak Forest, Illinois
  - Donald R. Graham, M.D., Springfield, Illinois
  - Alvaro G. Koch, M.D., Lexington, Kentucky
  - Shaban Faruqui, M.D., Baton Rouge, Louisiana
  - Robert M. Be, M.D., Baton Rouge, Louisiana
  - Bal Raj Bhandari, M.D., Monroe, Louisiana
  - Luis A. Balart, M.D., New Orleans, Louisiana
  - Robert Perrillo, M.D., New Orleans, Louisiana
  - Michael Epstein, M.D., Annapolis, Maryland
  - Natarajan Ravendhran, M.D., Baltimore, Maryland
  - Mark Sulkowski, M.D., Baltimore, Maryland
  - Milton J. Koch, M.D., Silver Spring, Maryland
  - David N. Schwartz, M.D., Attleboro, Massachusetts
  - Nezam Afdhal, M.D., Boston, Massachusetts
  - Lawton Shick, M.D., Worcester, Massachusetts
  - Stuart C. Gordon, M.D., Detroit, Michigan
  - John B. Gross, M.D., Rochester, Minnesota
  - Jeffrey Rank, M.D., Saint Paul, Minnesota
  - Adrian Di Bisceglie, M.D., St Louis, Missouri
  - William C. Sloan, Florham Park, New Jersey
  - Rajendra Prasad Gupta, M.D., Trenton, New Jersey
  - David Eric Bernstein, M.D., Manhasset, New York
  - Ira M. Jacobson, M.D., New York, New York
  - Douglas T. Dieterich, M.D., New York, New York
  - Robert Reindollar, M.D., Charlotte, North Carolina
  - Andrew Muir, M.D., Durham, North Carolina
  - John E. Poulous, M.D., Fayetteville, North Carolina
  - Mark E. Jonas, M.D., Cincinnati, Ohio
  - Harvey A. Tatum, M.D., Tulsa, Oklahoma
  - George Koval, M.D., Portland, Oregon
  - Jill P. Smith, M.D., Hershey, Pennsylvania
  - Victor Araya, M.D., Philadelphia, Pennsylvania
  - Peter J. Molloy, M.D., Pittsburgh, Pennsylvania
  - James Scott Strohecker, M.D., Columbia, South Carolina
  - Lawrence D. Wruble, M.D., Memphis, Tennessee
  - Ronald Pruitt, M.D., Nashville, Tennessee
  - Gary L. Davis, M.D., Dallas, Texas
  - William M. Lee, M.D., Dallas, Texas
  - George G. Burnazian, M.D., Houston, Texas
  - Rise Stribling, M.D., Houston, Texas
  - Eric J. Lawitz, M.D., San Antonio, Texas
  - Daniel Pambianco, M.D., Charlottesville, Virginia
  - Vinod Rustgi, M.D., Fairfax, Virginia
  - Mitchell Shiffman, M.D., Richmond, Virginia
  - Robert A. Wohlman, M.D., Bellevue, Washington
  - Robert L. Carithers, M.D., Seattle, Washington
  - David Winters McEniry, M.D., Tacoma, Washington
  - Michael F. Lyons II, M.D., Tacoma, Washington

REFERENCES:
- [Derived] Rustgi VK, Lee WM, Lawitz E, Gordon SC, Afdhal N, Poordad F, Bonkovsky HL, Bengtsson L, Chandorkar G, Harding M, McNair L, Aalyson M, Alam J, Kauffman R, Gharakhanian S, McHutchison JG; MErimepodib TRiple cOmbination Study Group. Merimepodib, pegylated interferon, and ribavirin in genotype 1 chronic hepatitis C pegylated interferon and ribavirin nonresponders. Hepatology. 2009 Dec;50(6):1719-26. doi: 10.1002/hep.23204. PMID 19852040